CLINICAL TRIAL: NCT01911689
Title: Magnetic Resonance Imaging Study of Acute Pancreatitis
Status: Completed | Type: Observational
Sponsor: Afﬁliated Hospital of North Sichuan Medical College (Other)
Responsible Party: Sponsor
Other Study IDs: SKLMC-2013-001
Record Dates: First submitted 2013-07-26; First posted 2013-07-30 (Estimated); Results first posted 2015-08-24 (Estimated); Last update posted 2015-08-24 (Estimated); Status verified 2014-11

CONDITIONS: Acute Pancreatitis
Keywords: pancreatitis; MRI; APACHEⅡ; T2*; T2 star
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- acute pancreatitis: acute pancreatitis group：(a) acute onset of abdominal pain; (b) pancreatitis at first onset; (c) three-fold elevated amylase or lipase, excluding other causes of elevated enzymes; and (5) abdominal MR examination.
- controlgroup: normal control group：without pancreatic disorders.The exclusion criteria in this study were as follows: (a) inability to cooperate when MR imaging was performed; (b) a history of chronic pancreatitis; (c) AP due to pancreatic carcinoma; (d) hypoproteinemia; and (e) with hypoproteinemia and other peritoneal/ retroperitoneal infection diseases ;(f) with iron deposition disorder (e.g. diabetes or blood system diseases).

SUMMARY:
To quantitatively analyze the T2* values of the head, body, and tail of normal pancreas, and observe the value of GRE T2*-weighted MRI in the diagnosis of acute pancreatitis and the relationship between the T2* value and the severity of AP.

DETAILED DESCRIPTION:
1. We design a prospective study about "Magetic Resonance Imaging Study of Acute Pancreatitis".
2. We apply for an account and register our study on the clinicalTrials.
3. In patients with acute pancreatitis, imaging is recommended to confirm the clinical diagnosis, investigate the etiology, and grade the severity of the disease . MR had the excellent resolution of soft tissue，and it has earned an ever more important role in the diagnosis of AP. With the continuous development of MR scanning techniques, the sequence of a multi-echo gradient recalled echo (GRE) T2*-weighted imaging (T2*WI), which acquires a spin echo signal, T2* relaxation acquires a gradient echo signal, is a relatively new MRI technique. The sequence of a GRE T2*WI requires high uniformity of the magnetic field, plus it can provide the T2* value, which can indirectly reflect changes in tissue biochemical components, thus it can be used for the early diagnosis quantitative diagnosis of some diseases .
4. This calculation process for T2* value is completed using post-processing software on the workstation(Advantage workstation 4.4; GE Halthcare) directly after scanning.
5. AP is a process of inflammation diffusion, in which cell edema will lead to hydrogen proton increase. In the inflammatory exudation process, T2* value will change. So we conduct our research. In this study, we will observe pancreas in the normal pancreas and AP, and discuss the relationship between T2* value and that of AP graded by the MR severity index (MRSI) and Acute Physiology And Chronic Healthy Evaluation II (APACHE II) scores.
6. However, until now, there is no research on the sequence applied in the patients with AP.

ELIGIBILITY:
Inclusion Criteria:

* acute onset of abdominal pain;
* pancreatitis at first onset;
* three-fold elevated amylase or lipase, excluding other causes of elevated enzymes; and
* abdominal MR examination.

Exclusion Criteria:

* inability to cooperate when MR imaging was performed;
* a history of chronic pancreatitis;
* AP due to pancreatic carcinoma;
* hypoproteinemia;
* with hypoproteinemia and other peritoneal/ retroperitoneal infection diseases ;
* with iron deposition disorder (e.g. diabetes or blood system diseases).

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with AP admitted to our institution between August 2013 and March 2015 were considered for inclusion in this study. The inclusion criteria for patients in this study were as follows: (a) acute onset of abdominal pain; (b) pancreatitis at first onset; (c) three-fold elevated amylase or lipase, excluding other causes of elevated enzymes; and (d) abdominal MR examination.
Sampling Method: Probability Sample
Enrollment: 168 (Actual)
Dates: Start 2013-08; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: zhang x ming, PHD, Study Chair — Afﬁliated Hospital of North Sichuan Medical College
Locations (1):
- Afﬁliated Hospital of North Sichuan Medical College, Nanchong, Sichuan, China

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with AP admitted to our institution between August 2013 and March 2015 were recruited in this study.
Pre-assignment Details: Patients with iron deposition disorder or chroic blood system diseases should be excluded in this study, because these diseases can lead to the change of the T2* value.
Period: Overall Study
Arm/Group | Acute Pancreatitis | Controlgroup
Started | 117 | 51
Completed | 117 | 51
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Acute Pancreatitis: All AP patients underwent the MRI scan within three days after admission. All MRI examinations were performed with a 3.0T scanner (Discovery MR 750; GE Medical Systems, Milwaukee, Wis) in the supine position.
- Controlgroup: All MRI examinations were performed with a 3.0T scanner (Discovery MR 750; GE Medical Systems, Milwaukee, Wis) in the supine position.
- Total: Total of all reporting groups
Arm/Group | Acute Pancreatitis | Controlgroup | Total
Number analyzed (Participants) | 117 | 51 | 168
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.41 (15.55) | 50.90 (17.83) | 50.56 (16.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 20 | 65
  Male | 72 | 31 | 103
Region of Enrollment [Number; unit: participants]
  China | 117 | 51 | 168

OUTCOME MEASURES:

1. Primary Outcome: The T2* Values in the Diagnosis of AP
Description: Compare the difference of the T2* value between the AP group and the control group.
Time Frame: 1 year
Population: compare T2* value between the AP group and the control group using independent sample t test
Measure: Mean (Standard Deviation); unit: ms
Groups:
- Acute Pancreatitis: T2* value of AP group is mean T2* values of the head, body and tail of pancreas respectively (If AP with necrosis, measureing the corresponding to the area with no necrosis).The AP group:(a) acute onset of abdominal pain; (b) pancreatitis at first onset; (c) three-fold elevated amylase or lipase, excluding other causes of elevated enzymes; and (5) abdominal MR examination
- Control Group: T2* value of control group is mean T2* values of the head, body and tail of pancreas respectively.The control group:without pancreatic disorders
Arm/Group | Acute Pancreatitis | Control Group
Number analyzed (Participants) | 117 | 51
ms | 25.86 (4.90) | 21.06 (2.64)
Statistical Analysis 1: Comparison: Acute Pancreatitis vs Control Group; The independent T test was used to determine the differences for the T2* value between the Control group and AP group; Test type: Superiority or Other; p < 0.01, t-test, 2 sided

2. Secondary Outcome: The Difference of T2* Value Between the Edematous AP and Necrotizing AP
Description: Compare the difference of the T2* value between the edematous AP group and necrotizing AP group
Time Frame: 1 year
Population: compare the difference of T2* value between the edematous AP and necrotizing AP
Measure: Mean (Standard Deviation); unit: ms
Groups:
- Edematous AP: T2* value of edematous AP
- Necrotizing AP: T2* value of necrotizing AP
Arm/Group | Edematous AP | Necrotizing AP
Number analyzed (Participants) | 93 | 24
ms | 25.28 (4.56) | 28.10 (5.59)
Statistical Analysis 1: Comparison: Edematous AP vs Necrotizing AP; The independent T test was used to determine the differences for the T2* value between the edematous AP and necrotizing AP; Test type: Superiority or Other; p = 0.05, t-test, 2 sided

3. Secondary Outcome: The T2* Value in Different Severity of AP According to MRSI
Description: AP was graded as mild (0-3 points), moderate (4-6 points) or severe (7-10 points), according to the MR-severity index (MRSI) which was derived from the CT-severity index .
Time Frame: 1 year
Population: AP was graded as mild (0-3 points), moderate (4-6 points) or severe (7-10 points), according to the MR-severity index (MRSI) which was derived from the CT-severity index .
Measure: Mean (Standard Deviation); unit: ms
Groups:
- Mild AP: Mild AP was defined as 0-3 points according to MRSI.
- Moderate AP: Moderate AP was defined as 4-6 points according to MRSI.
- Severe AP: Severe AP was defined as 7-10 points according to MRSI.
Arm/Group | Mild AP | Moderate AP | Severe AP
Number analyzed (Participants) | 41 | 69 | 7
ms | 24.08 (4.41) | 26.49 (4.91) | 29.99 (3.83)
Statistical Analysis 1: Comparison: Mild AP vs Moderate AP vs Severe AP; Analysis of variance (ANOVA) was used to assess the differences in the T2* value between the mild, moderate, and severe AP groups according to the MRSI score; Test type: Superiority or Other; p < 0.01, ANOVA
Statistical Analysis 2: Comparison: Mild AP vs Moderate AP; compare the T2* value in the mild and moderate AP according to MRSI; Test type: Superiority or Other; p = 0.0111, t-test, 2 sided
Statistical Analysis 3: Comparison: Mild AP vs Severe AP; compare the T2* value between the mild and severe AP; Test type: Superiority or Other; p = 0.002, t-test, 2 sided
Statistical Analysis 4: Comparison: Moderate AP vs Severe AP; compare the T2* value between the moderate and severe AP according to MRSI; Test type: Superiority or Other; p = 0.071, t-test, 2 sided

4. Secondary Outcome: The Relationship Between the T2* Value and the Severity of AP According to Apache II
Description: In clinical practice, the physician usually used the APACHE II to evaluate the severity of acute pancreatitis. AP was graded as mild (0-7 points) and severe AP (≥8 points) according to the APACHE II scoring system.
Time Frame: 1 year
Population: Indengpent T test
Measure: Mean (Standard Deviation); unit: ms
Groups:
- Mild AP: Mild AP was graded as the Apache II score < 7 points.
- Severe AP: Severe AP was graded as the Apache II score ≥8 points.
Arm/Group | Mild AP | Severe AP
Number analyzed (Participants) | 89 | 28
ms | 25.73 (4.80) | 26.25 (5.26)
Statistical Analysis 1: Comparison: Mild AP vs Severe AP; Test type: Superiority or Other; p = 0.629, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 6 months
Groups:
- Acute Pancreatitis; Controlgroup: Not Including Serious
Arm/Group | Acute Pancreatitis | Controlgroup
Serious Adverse Events (participants affected / at risk) | 0/117 | 0/51
Other Adverse Events (participants affected / at risk) | 0/117 | 0/51

LIMITATIONS AND CAVEATS:
Some diseases, such as chronic anemia, diabetes, etc., may lead to iron deposition in pancreas and may lead to change the T2* value.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes